CLINICAL TRIAL: NCT01511419
Title: Reactogenicity, Safety and Immunogenicity of a Live Monovalent A/17/Mallard/Netherlands/00/95 (H7N3) Influenza Vaccine
Brief Title: Safety Trial of Live Attenuated Influenza (H7N3) Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Ministry of Health, Russian Federation (Other Government); Research Institute of Influenza, Russia (Other); Institute of Experimental Medicine, Russia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LAIV-H7N3-01
Record Dates: First submitted 2012-01-05; First posted 2012-01-18 (Estimated); Results first posted 2019-04-22 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-01

CONDITIONS: Influenza; Avian Influenza
Keywords: Influenza; Vaccine; Pandemic; H7N3
MeSH Terms: conditions — Influenza, Human; Influenza in Birds

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LAIV H7N3 (Experimental): Test drug/agent: Live-attenuated A/17/mallard/Netherlands/00/95 influenza vaccine (LAIV H7N3) grown in embryonated chicken eggs.
  Name of active ingredient(s): Live-attenuated A/17/mallard/Netherlands/00/95 influenza vaccine.
  Dose: ≥7.5 log egg infectious dose (EID) 50/0.5 ml dose; 0.25 ml/nare.
  Route of administration: Intranasal aerosol.
  Duration of treatment: Two doses were delivered, one on Day 0 and one on Day 28.
  Interventions: Biological: LAIV H7N3
- Placebo (Placebo Comparator): Reference drug: Placebo; saline inoculated in embryonated chicken eggs and subsequently prepared in the same way as test vaccine.
  Dose: 0.5 ml; 0.25 ml/nare
  Route of administration: Intranasal aerosol
  Duration of treatment: Two doses were delivered, one on Day 0 and one on Day 28
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: LAIV H7N3 — 2 doses of vaccine
  Other Names: A/17/mallard/Netherlands/00/95 (H7N3)
  Arms: LAIV H7N3
Biological: placebo — 2 doses of placebo
  Arms: Placebo

SUMMARY:
The study hypothesis is that two doses of cold-adapted, live monovalent A/17/mallard/Netherlands/00/95 (H7N3) influenza vaccine will be safe and immunogenic in healthy adults.

DETAILED DESCRIPTION:
This is a phase I, double-blind, individually-randomized (3:1, vaccine:placebo), controlled trial with two groups, LAIV H7N3 and matched placebo. Healthy male and female adults 18 through 49 years of age will be invited to participate. For feasibility reasons and in order for an independent Safety Monitoring Committee (SMC) to review safety data in a small group of subjects initially, the total cohort of 40 subjects will be enrolled in two sub-cohorts: one cohort of 12 subjects, randomized at 3:1 (9 vaccine and 3 placebo), followed two weeks later by a second cohort of 28 subjects randomized at 3:1 (21 vaccine and 7 placebo). After all 12 volunteers of the first sub-cohort have been observed for the first isolation period (Day 1 to Day 7), an interim safety review will be performed by the SMC. The SMC will review all adverse events (AEs), including clinical laboratory evaluations (pre- and post-vaccination) and shedding data, for all subjects and will advise if the volunteers of the first sub-cohort may receive dose two of study vaccine or placebo and if the additional 28 volunteers of the second sub-cohort may be enrolled into the study. As for the first sub-cohort, the SMC will also review all safety data for the second sub-cohort and for the entire participant population of the trial. For each sub-cohort, the procedures and timelines are here summarized.

On the day of first screening, about 7 days (between 4 and 14 days) prior to administration of dose one of study vaccine or placebo, subjects will be screened for eligibility through medical history review, physical examination, testing for serologic evidence of chronic viral infection [human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV), with proper pre- and post-test counseling], routine biochemical and hematological blood tests and urinalysis by dipstick.

Subject screening for eligibility will continue and be completed on the second screening day (S2). This second screening day will occur the same day as scheduled admission to the isolation unit and administration of study vaccine or placebo (Day 0). Women will undergo pregnancy tests using urine samples. All subjects will undergo an ear, nose and throat (ENT) examination. Fully eligible subjects will be admitted to the isolation unit. At that time, nasal swab, nasal wick, and blood specimens will be collected for virologic and immunological testing prior to administration of study vaccine or placebo. Blood and urine specimens will be again collected for routine biochemical and hematological blood tests and urinalysis by dipstick; these results will serve to define baseline status for subject prior to receipt of study vaccine or placebo but will not be used for screening purposes. Subjects will be unaware of which allocation, LAIV H7N3 or matched placebo, is received; study vaccine and placebo will be masked. Subjects will be carefully monitored for adverse reactions while in the isolation unit.

All subjects will remain in the isolation unit for at least 7 days after receipt of study vaccine or placebo. Nasal swabs will be collected daily while subjects are in isolation to test for presence of influenza virus shed in the nasal passage. Any subject exhibiting conjunctivitis will also have a conjunctival swab collected on the day of appearance of the sign. Any subject exhibiting influenza A virus shedding, as determined by real-time reverse transcriptase polymerase chain reaction (RT-PCR) positivity on a nasal swab specimen, in the 2 days prior to each planned discharge day after each dose (Days 6 or 7 or Days 34 or 35) will be kept in the isolation until PCR-diagnosis results confirm that no influenza virus is present in a tested clinical specimen for at least two consecutive days. Any subject still exhibiting evidence of influenza virus shedding in a nasal swab on Days 6 or 7 or Days 34 or 35 post-administration with each dose might be placed on influenza antiviral (oseltamivir) treatment at the standard dose for treatment of 75 milligrams (mg) twice a day for a course of 5 days.

After discharge from the isolation unit, subjects will complete diary cards for AEs and use of concomitant medications. Subjects will return to the isolation unit at four weeks (Day 28) after administration of dose one of study vaccine or placebo. At that time, similar procedures will be used for admittance to the isolation unit, for receipt of dose two of study vaccine or placebo and for isolation and follow-up, with the additional procedure of review of interim histories (and diary cards) since first discharge after dose one.

After second discharge from the isolation unit, subjects will again complete diary cards for AEs and use of concomitant medications. Subjects will then return to the study center at four weeks (Day 56) after administration of dose two of study vaccine or placebo for their final study visit. Interim histories (and diary cards) will again be reviewed and final blood and nasal wick specimens will be collected. Women will also undergo a final pregnancy screen. Subjects will complete the study at this time.

For assessment of safety, subjects will be observed for two hours after each administration of study vaccine or placebo. Twice daily (early morning and late afternoon) examination will be also used to assess reactions for 7 days after each administration of study vaccine or placebo. ENT examination will also occur once per day on Days 7, 28, 35 and 56. Subjects will complete diary cards for unsolicited AEs from the day of each discharge until return to the isolation unit for dose two (at Day 28) or until return to the study center for the final study visit at four weeks post dose two (at Day 56). To assess safety, blood and urine specimens will also be collected on days 7, 28 (prior to administration of dose two of study vaccine or placebo), 35 and 56, for testing by routine biochemical and hematological blood tests and by urinalysis by dipstick.

For the evaluation of mucosal immunoglobulin A (IgA) antibody, nasal wick specimens will be collected on Day 0 (prior to administration of dose one of study vaccine or placebo), on Day 28 (prior to administration of dose two of study vaccine or placebo) and on Day 56. For the evaluation of serum antibodies (by hemagglutination inhibition [HAI], microneutralization and IgA and immunoglobulin G [IgG] EIA), serum specimens will be collected on Day 0 (prior to administration of dose one of study vaccine or placebo), on Day 28 (prior to administration of dose two of study vaccine or placebo) and on Day 56. To study virus infectivity (by isolation in chicken embryos) and stability (by molecular sequencing of any isolated virus), nasal swab specimens will be taken on Days 1, 2, 3, 5, 7, 29, and 31. To assess priming and stimulation of cytotoxic T lymphocytes and other cytokine indicators, whole blood for isolation of peripheral blood mononuclear cells (PBMCs) will be collected on Days 0 (prior to administration of dose one of study vaccine or placebo), on Day 28 (prior to administration of dose two of study vaccine or placebo) and on Day 56.

ELIGIBILITY:
Inclusion Criteria:

* Legal male or female adult 18 through 49 years of age at the enrollment visit.
* Literate and willing to provide written informed consent.
* Free of obvious health problems, as established by the medical history and screening evaluations, including physical examination.
* Capable and willing to complete diary cards and willing to return for all follow-up visits
* Willing to comply with the rules of the isolation unit (including willing and able to take oseltamivir influenza antiviral medication, should that be recommended by a study physician).
* For females, willing to take reliable birth control measures throughout the entire period of participation in the study.

Exclusion Criteria:

* Participation in another clinical trial involving any therapy within the previous three months or planned enrollment in such a trial during the period of this study.
* Receipt of any non-study vaccine within four weeks prior to enrollment or refusal to postpone receipt of such vaccines until four weeks after study completion.
* Practice of nasal irrigation on a regular basis within the past six months or has engaged in nasal irrigation within two weeks prior to enrollment.
* Recent history of frequent nose bleeds (>5 within the past year).
* Clinically relevant abnormal paranasal anatomy.
* Recent history (within the past month) of rhino or sinus surgery, or surgery for any traumatic injury of the nose.
* Current or recent (within two weeks of enrollment) acute respiratory illness with or without fever.
* Other acute illness at the time of study enrollment.
* Receipt of immune globulin or other blood products within three months prior to study enrollment or planned receipt of such products during the period of subject participation in the study.
* Chronic administration (defined as more than 14 consecutively-prescribed days) of immunosuppressants or other immune-modulating therapy within six months prior to study enrollment. (For corticosteroids, this means prednisone or equivalent, >=0.5 mg per kg per day; topical steroids are allowed, exclusive of nasal.)
* Participation in any previous trial of any H5 or H7 containing influenza vaccine.
* History of asthma.
* Hypersensitivity after previous administration of any influenza vaccine.
* History of wheezing after past receipt of any live influenza vaccine.
* Other AE following immunization, at least possibly related to previous receipt of any influenza vaccine.
* Suspected or known hypersensitivity to any of the study vaccine components, including chicken or egg protein.
* Seasonal (autumnal) hypersensitivity to the natural environment.
* Acute or chronic clinically significant pulmonary, cardiovascular, hepatic, metabolic, neurologic, psychiatric or renal functional abnormality, as determined by medical history, physical examination or clinical laboratory screening tests, which in the opinion of the investigator, might interfere with the study objectives. Subjects with physical examination findings or clinical laboratory screening results which would be graded 2 or higher on the AE severity grading scale will be excluded from entry into the study and will be excluded from receipt of dose two of study vaccine or placebo.
* History of leukemia or any other blood or solid organ cancer.
* History of thrombocytopenic purpura or known bleeding disorder.
* History of seizures.
* Known or suspected immunosuppressive or immunodeficient condition of any kind, including HIV infection.
* Known chronic HBV or HCV infection.
* Known tuberculosis infection or evidence of previous tuberculosis exposure.
* History of chronic alcohol abuse and/or illegal drug use.
* Claustrophobia or sociophobia.
* Pregnancy or lactation. (A negative pregnancy test will be required before administration of study vaccine or placebo for all women of childbearing potential.)
* Any condition that, in the opinion of the investigator, would increase the health risk to the subject if he/she participates in the study or would interfere with the evaluation of the study objectives.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oleg I Kiselev, MD, PhD, DSc, Principal Investigator — Research Institute of Influenza; Larisa G Rudenko, MD, PhD, DSc, Study Director — Institute of Experimental Medicine; Kathleen M Neuzil, MD, MPH, Study Director — PATH Vaccine Solutions; Igor Victorevich, Study Director — Microgen
Locations (1):
- Research Institute of Influenza, Saint Petersburg, Russia

REFERENCES:
- [Derived] Kiseleva I, Dubrovina I, Fedorova E, Larionova N, Isakova-Sivak I, Bazhenova E, Pisareva M, Kuznetsova V, Flores J, Rudenko L. Genetic stability of live attenuated vaccines against potentially pandemic influenza viruses. Vaccine. 2015 Dec 8;33(49):7008-14. doi: 10.1016/j.vaccine.2015.09.050. Epub 2015 Oct 2. PMID 26432909
- [Derived] Rudenko L, Kiseleva I, Naykhin AN, Erofeeva M, Stukova M, Donina S, Petukhova G, Pisareva M, Krivitskaya V, Grudinin M, Buzitskaya Z, Isakova-Sivak I, Kuznetsova S, Larionova N, Desheva J, Dubrovina I, Nikiforova A, Victor JC, Neuzil K, Flores J, Tsvetnitsky V, Kiselev O. Assessment of human immune responses to H7 avian influenza virus of pandemic potential: results from a placebo-controlled, randomized double-blind phase I study of live attenuated H7N3 influenza vaccine. PLoS One. 2014 Feb 12;9(2):e87962. doi: 10.1371/journal.pone.0087962. eCollection 2014. PMID 24533064

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Reference drug: Placebo; saline inoculated in embryonated chicken eggs and subsequently prepared in the same way as test vaccine.
  Dose: 0.5 ml; 0.25 ml/nare
  Route of administration: Intranasal aerosol
  Duration of treatment: Two doses were delivered, one on Day 0 and one on Day 28
  placebo: 2 doses of placebo
Period: Dose 1
Arm/Group | LAIV H7N3 | Placebo
Started | 30 | 10
Completed | 30 | 10
Not Completed | 0 | 0
Period: Dose 2
Arm/Group | LAIV H7N3 | Placebo
Started | 30 | 10
Completed | 29 | 10
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- LAIV H7N3: Test drug/agent: Live-attenuated A/17/mallard/Netherlands/00/95 influenza vaccine (LAIV H7N3) grown in embryonated chicken eggs.
  Name of active ingredient(s): Live-attenuated A/17/mallard/Netherlands/00/95 influenza vaccine.
  Dose: ≥7.5 log EID50/0.5 ml dose; 0.25 ml/nare.
  Route of administration: Intranasal aerosol.
  Duration of treatment: Two doses were delivered, one on Day 0 and one on Day 28.
  LAIV H7N3: 2 doses of vaccine
- Total: Total of all reporting groups
Arm/Group | LAIV H7N3 | Placebo | Total
Number analyzed (Participants) | 30 | 10 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.1 (10.3) | 38.5 (9.7) | 32.2 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 4 | 19
  Male | 15 | 6 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Immediate Reactions
Description: From administration of any dose, immediate reaction measured as observed by study staff or reported by the subject to study staff in case of an anaphylactic reaction.
Time Frame: 2 hours post-administration on Days 0 and 28
Population: Intent-to-treat (ITT) population
Measure: Count of Participants; unit: Participants
Groups:
- LAIV H7N3: Dose 1 (Day 0); LAIV H7N3: Dose 2 (Day 28): Test drug/agent: Live-attenuated A/17/mallard/Netherlands/00/95 influenza vaccine (LAIV H7N3) grown in embryonated chicken eggs.
  Name of active ingredient(s): Live-attenuated A/17/mallard/Netherlands/00/95 influenza vaccine.
  Dose: ≥7.5 log EID50/0.5 ml dose; 0.25 ml/nare.
  Route of administration: Intranasal aerosol.
- Placebo: Dose 1 (Day 0); Placebo: Dose 2 (Day 28): Reference drug: Placebo; saline inoculated in embryonated chicken eggs and subsequently prepared in the same way as test vaccine.
  Dose: 0.5 ml; 0.25 ml/nare
  Route of administration: Intranasal aerosol
Arm/Group | LAIV H7N3: Dose 1 (Day 0) | Placebo: Dose 1 (Day 0) | LAIV H7N3: Dose 2 (Day 28) | Placebo: Dose 2 (Day 28)
Number analyzed (Participants) | 30 | 10 | 29 | 10
Participants
  Immediate reaction | 0 | 0 | 0 | 0
  No immediate reaction | 30 | 10 | 29 | 10

2. Primary Outcome: Adverse Events Associated With Intranasal Vaccination
Description: From solicited local and systemic reactions
Time Frame: Greater than 2 hours through 7 days following any dose
Population: Intent-To-Treat (ITT) Population
Measure: Count of Participants; unit: Participants
Groups:
- LAIV H7N3: Dose 1; LAIV H7N3: Dose 2: Test drug/agent: Live-attenuated A/17/mallard/Netherlands/00/95 influenza vaccine (LAIV H7N3) grown in embryonated chicken eggs.
  Name of active ingredient(s): Live-attenuated A/17/mallard/Netherlands/00/95 influenza vaccine.
  Dose: ≥7.5 log EID50/0.5 ml dose; 0.25 ml/nare.
  Route of administration: Intranasal aerosol.
- Placebo: Dose 1; Placebo: Dose 2: Reference drug: Placebo; saline inoculated in embryonated chicken eggs and subsequently prepared in the same way as test vaccine.
  Dose: 0.5 ml; 0.25 ml/nare
  Route of administration: Intranasal aerosol
Arm/Group | LAIV H7N3: Dose 1 | Placebo: Dose 1 | LAIV H7N3: Dose 2 | Placebo: Dose 2
Number analyzed (Participants) | 30 | 10 | 29 | 10
Participants
  Any local or systemic reaction | 11 | 4 | 5 | 1
  No local or systemic reaction | 19 | 6 | 24 | 9

3. Primary Outcome: All Other Adverse Events
Description: Including unsolicited events and abnormal laboratory findings
Time Frame: 7 days following any dose
Population: Total events among Intent-To-Treat (ITT) Population
Measure: Count of Units; unit: adverse events
Units Other Than Participants: adverse events
Arm/Group | LAIV H7N3: Dose 1 | Placebo: Dose 1 | LAIV H7N3: Dose 2 | Placebo: Dose 2
Number analyzed (Participants) | 30 | 10 | 29 | 10
Number analyzed (adverse events) | 44 | 6 | 90 | 21
adverse events
  Unrelated | 40 | 6 | 84 | 20
  Related | 4 | 0 | 6 | 1

4. Primary Outcome: Participants With Serious Adverse Events (SAEs)
Description: Including abnormal laboratory findings
Time Frame: Within 4 weeks of receipt of any dose
Population: Intent-To-Treat (ITT) Population
Measure: Count of Participants; unit: Participants
Arm/Group | LAIV H7N3: Dose 1 | Placebo: Dose 1 | LAIV H7N3: Dose 2 | Placebo: Dose 2
Number analyzed (Participants) | 30 | 10 | 29 | 10
Participants
  Any serious adverse event | 0 | 0 | 0 | 0
  No serious adverse event | 30 | 10 | 29 | 10

5. Secondary Outcome: Number/Percentage of Subjects With Seroconversion for Serum Hemagglutination Inhibition (HAI)
Description: Seroconversion was defined as at least a four-fold rise after each dose from baseline or as the mean titer after each dose
Time Frame: 28 days (Dose 1) and 56 days (Dose 2)
Population: Per-Protocol (PP) Population
Measure: Count of Participants; unit: Participants
Arm/Group | LAIV H7N3: Dose 1 | Placebo: Dose 1 | LAIV H7N3: Dose 2 | Placebo: Dose 2
Number analyzed (Participants) | 29 | 10 | 29 | 10
Participants
  Seroconversion | 3 | 0 | 9 | 0
  No seroconversion | 26 | 10 | 20 | 10

6. Secondary Outcome: Number/Percentage of Subjects With Serum Neutralizing Antibodies
Description: Measured using microneutralization assay. Seroconversion was defined as at least a four-fold rise after each dose from baseline or as the mean titer after each dose
Time Frame: 28 days (Dose 1) and 56 days (Dose 2)
Population: Per-Protocol (PP) Population
Measure: Count of Participants; unit: Participants
Arm/Group | LAIV H7N3: Dose 1 | Placebo: Dose 1 | LAIV H7N3: Dose 2 | Placebo: Dose 2
Number analyzed (Participants) | 29 | 10 | 29 | 10
Participants
  Seroconversion | 5 | 0 | 12 | 0
  No seroconversion | 24 | 10 | 17 | 10

7. Secondary Outcome: Number/Percentage of Subjects With Seroconversion for Serum Immunoglobulin A (IgA)
Description: Measured by enzyme-linked immunoassay (EIA). Seroconversion was defined as at least a four-fold rise after each dose from baseline or as the mean titer after each dose
Time Frame: 28 days (Dose 1) and 56 days (Dose 2)
Population: Per-Protocol (PP) Population
Measure: Count of Participants; unit: Participants
Arm/Group | LAIV H7N3: Dose 1 | Placebo: Dose 1 | LAIV H7N3: Dose 2 | Placebo: Dose 2
Number analyzed (Participants) | 29 | 10 | 29 | 10
Participants
  Seroconversion | 3 | 0 | 8 | 0
  No seroconversion | 26 | 10 | 21 | 10

8. Secondary Outcome: Number/Percentage of Subjects With Seroconversion for Serum Immunoglobulin G (IgG)
Description: as for outcome 7
Time Frame: 28 days (Dose 1) and 56 days (Dose 2)
Population: Per-Protocol (PP) Population
Measure: Count of Participants; unit: Participants
Arm/Group | LAIV H7N3: Dose 1 | Placebo: Dose 1 | LAIV H7N3: Dose 2 | Placebo: Dose 2
Number analyzed (Participants) | 29 | 10 | 29 | 10
Participants
  Seroconversion | 1 | 0 | 3 | 0
  No seroconversion | 28 | 10 | 26 | 10

9. Secondary Outcome: Number/Percentage of Subjects With Seroconversion for Mucosal IgA
Description: From nasal wick specimen. Seroconversion was defined as at least a four-fold rise after each dose from baseline or as the mean titer after each dose
Time Frame: 28 days (Dose 1) and 56 days (Dose 2)
Population: Per-Protocol (PP) Population
Measure: Count of Participants; unit: Participants
Arm/Group | LAIV H7N3: Dose 1 | Placebo: Dose 1 | LAIV H7N3: Dose 2 | Placebo: Dose 2
Number analyzed (Participants) | 29 | 10 | 29 | 10
Participants
  Seroconversion | 12 | 1 | 12 | 1
  No seroconversion | 17 | 9 | 17 | 9

10. Secondary Outcome: Geometric Mean Titers (GMTs) for Serum Hemagglutination Inhibition (HAI) Antibodies (4 Haemagglutinating Units of H7N3)
Description: HAI test was performed by standard procedure with human red blood cells utilizing either 4 haemagglutinating units (HAU) of H7N3.
Time Frame: 0 days, 28 days (Dose 1) and 56 days (Dose 2)
Population: Per-Protocol (PP) Population
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | LAIV H7N3 | Placebo
Number analyzed (Participants) | 29 | 10
titers
  Day 0 | 2.8 [2.5 to 3.1] | 3.3 [2.3 to 4.7]
  Day 28 | 3.5 [2.8 to 4.4] | 3.3 [2.3 to 4.7]
  Day 56 | 4.7 [3.5 to 6.1] | 3.5 [2.5 to 5.0]

11. Secondary Outcome: Geometric Mean Titers (GMTs) for Serum Hemagglutination Inhibition (HAI) Antibodies (2 Haemagglutinating Units of H7N3)
Description: HAI test was performed by standard procedure with human red blood cells utilizing 2 haemagglutinating units (HAU) of H7N3.
Time Frame: 0 days, 28 days (Dose 1) and 56 days (Dose 2)
Population: Per-Protocol (PP) population
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | LAIV H7N3 | Placebo
Number analyzed (Participants) | 29 | 10
titer
  Day 0 | 3.0 [2.6 to 3.5] | 4.1 [2.7 to 6.1]
  Day 28 | 5.5 [4.2 to 7.2] | 4.1 [2.7 to 6.1]
  Day 56 | 7 [5.2 to 9.4] | 4.7 [2.8 to 7.6]

12. Secondary Outcome: Geometric Mean Titers (GMTs) for Serum Neutralizing Antibodies
Description: Measured by microneutralization assay
Time Frame: 0 days, 28 days (Dose 1) and 56 days (Dose 2)
Population: Per-Protocol (PP) population
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | LAIV H7N3 | Placebo
Number analyzed (Participants) | 29 | 10
titer
  Day 0 | 4.2 [3.5 to 5.1] | 4.4 [2.8 to 6.9]
  Day 28 | 6.2 [4.5 to 8.5] | 4.4 [2.8 to 6.9]
  Day 56 | 12.4 [8.2 to 18.7] | 5.0 [3.1 to 8.0]

13. Secondary Outcome: Number/Percentage of Vaccinated Subjects Shedding Virus After First Dose
Description: Detected by real-time reverse transcriptase polymerase chain reaction (rRTPCR) in nasal swabs or conjunctival swabs or by isolation in chicken embryos.
Time Frame: Days 1, 2, 3 & 4
Population: Intent-To-Treat (ITT) Population
Measure: Count of Participants; unit: Participants
Groups:
- Day 1; Day 2; Day 3; Day 4: LAIV H7N3 Arm
Arm/Group | Day 1 | Day 2 | Day 3 | Day 4
Number analyzed (Participants) | 30 | 30 | 30 | 30
Participants
  Shedding | 18 | 3 | 1 | 0
  No shedding | 12 | 27 | 29 | 30

14. Secondary Outcome: Number/Percentage of Subjects Shedding Virus After Second Dose
Description: as for outcome 13
Time Frame: Day 29, 30, 31 and 32
Population: Per-Protocol (PP) Population
Measure: Count of Participants; unit: Participants
Groups:
- Day 29; Day 30; Day 31; Day 32: LAIV H7N3 Arm
Arm/Group | Day 29 | Day 30 | Day 31 | Day 32
Number analyzed (Participants) | 29 | 29 | 29 | 29
Participants
  Shedding | 14 | 2 | 1 | 0
  No shedding | 15 | 27 | 28 | 29

15. Other Pre Specified Outcome: Number/Percentage of Subjects Exhibiting CD4+ IFNγ+ Responses
Description: H7N3-specific T cell responses were examined in peripheral blood mononuclear cells (PBMCs) obtained from all the study subjects before vaccination (Day 0), 28 days after the first vaccination (Day 28) and 28 days after revaccination (Day 56). To calculate the frequency of virus-specific T cells we quantified all cells positive for IFNγ after in vitro stimulation with whole H7N3 virion.
  Increases in the antigen-specific CD4+T-cell levels exceeding 3 standard deviations from the levels in the mean of the placebo were considered positive responses.
Time Frame: Days 0, 28 & 56
Population: Per-Protocol (PP) population that received 2 doses of either vaccine or placebo
Measure: Count of Participants; unit: Participants
Groups:
- LAIV H7N3: Day 0 (After Dose 1); LAIV H7N3: Day 28 (Dose 2); LAIV H7N3: Day 56 (28 Days Past Dose 2): Test drug/agent: Live-attenuated A/17/mallard/Netherlands/00/95 influenza vaccine (LAIV H7N3) grown in embryonated chicken eggs.
  Name of active ingredient(s): Live-attenuated A/17/mallard/Netherlands/00/95 influenza vaccine.
  Dose: ≥7.5 log EID50/0.5 ml dose; 0.25 ml/nare.
  Route of administration: Intranasal aerosol.
- Placebo: Day 0 (After Dose 1); Placebo: Day 28 (Dose 2); Placebo: Day 56 (28 Days Past Dose 2): Reference drug: Placebo; saline inoculated in embryonated chicken eggs and subsequently prepared in the same way as test vaccine.
  Dose: 0.5 ml; 0.25 ml/nare
  Route of administration: Intranasal aerosol
Arm/Group | LAIV H7N3: Day 0 (After Dose 1) | Placebo: Day 0 (After Dose 1) | LAIV H7N3: Day 28 (Dose 2) | Placebo: Day 28 (Dose 2) | LAIV H7N3: Day 56 (28 Days Past Dose 2) | Placebo: Day 56 (28 Days Past Dose 2)
Number analyzed (Participants) | 29 | 10 | 29 | 10 | 29 | 10
Participants
  Positive response | 2 | 0 | 3 | 0 | 4 | 0
  No response | 27 | 10 | 26 | 10 | 25 | 10

16. Other Pre Specified Outcome: Number/Percentage of Subjects Exhibiting CD4+ IFNγ+ Central Memory T Cell Responses
Description: H7N3-specific T cell responses were examined in PBMCs obtained from all the study subjects before vaccination (Day 0), 28 days after the first vaccination (Day 28) and 28 days after revaccination (Day 56). To calculate the frequency of virus-specific T cells we quantified all cells positive for IFNγ after in vitro stimulation with whole H7N3 virion.
  Increases in the antigen-specific CD4+T-cell levels exceeding 3 standard deviations from the levels in the mean of the placebo were considered positive responses.
Time Frame: Days 0, 28 & 56
Population: Per-Protocol (PP) population that received 2 doses of either vaccine or placebo
Measure: Count of Participants; unit: Participants
Arm/Group | LAIV H7N3: Day 0 (After Dose 1) | Placebo: Day 0 (After Dose 1) | LAIV H7N3: Day 28 (Dose 2) | Placebo: Day 28 (Dose 2) | LAIV H7N3: Day 56 (28 Days Past Dose 2) | Placebo: Day 56 (28 Days Past Dose 2)
Number analyzed (Participants) | 29 | 10 | 29 | 10 | 29 | 10
Participants
  Positive response | 5 | 0 | 6 | 0 | 7 | 0
  No response | 24 | 10 | 23 | 10 | 22 | 10

17. Other Pre Specified Outcome: Number/Percentage of Subjects Exhibiting CD4+ IFNγ+ Effector Memory T Cell Responses
Description: as for outcome 16
Time Frame: Days 0, 28 & 56
Measure: Count of Participants; unit: Participants
Arm/Group | LAIV H7N3: Dose 1 (Day 0) | Placebo: Dose 1 (Day 0) | LAIV H7N3: Day 28 (Dose 2) | Placebo: Day 28 (Dose 2) | LAIV H7N3: Day 56 (28 Days Past Dose 2) | Placebo: Day 56 (28 Days Past Dose 2)
Number analyzed (Participants) | 29 | 10 | 29 | 10 | 29 | 10
Participants
  Positive response | 1 | 0 | 3 | 0 | 3 | 0
  No response | 28 | 10 | 26 | 10 | 26 | 10

18. Other Pre Specified Outcome: Number/Percentage of Subjects Exhibiting CD8+ IFNγ+ Responses
Description: as for outcome 16
Time Frame: Days 0, 28 & 56
Population: Per-Protocol (PP) population that received 2 doses of either vaccine or placebo
Measure: Count of Participants; unit: Participants
Arm/Group | LAIV H7N3: Dose 1 (Day 0) | Placebo: Dose 1 (Day 0) | LAIV H7N3: Day 28 (Dose 2) | Placebo: Day 28 (Dose 2) | LAIV H7N3: Day 56 (28 Days Past Dose 2) | Placebo: Day 56 (28 Days Past Dose 2)
Number analyzed (Participants) | 29 | 10 | 29 | 10 | 29 | 10
Participants
  Positive response | 0 | 0 | 5 | 0 | 5 | 0
  No response | 29 | 10 | 24 | 10 | 24 | 10

19. Other Pre Specified Outcome: Number/Percentage of Subjects Exhibiting CD8+ IFNγ+ Central Memory T Cell Responses
Description: as for outcome 16
Time Frame: Days 0, 28 & 56
Population: Per-Protocol (PP) population that received 2 doses of either vaccine or placebo
Measure: Count of Participants; unit: Participants
Arm/Group | LAIV H7N3: Dose 1 (Day 0) | Placebo: Dose 1 (Day 0) | LAIV H7N3: Day 28 (Dose 2) | Placebo: Day 28 (Dose 2) | LAIV H7N3: Day 56 (28 Days Past Dose 2) | Placebo: Day 56 (28 Days Past Dose 2)
Number analyzed (Participants) | 29 | 10 | 29 | 10 | 29 | 10
Participants
  Positive response | 1 | 0 | 6 | 0 | 6 | 0
  No response | 28 | 10 | 23 | 10 | 23 | 10

20. Other Pre Specified Outcome: Number/Percentage of Subjects Exhibiting CD8+ IFNγ+ Effector Memory T Cell Responses
Description: as for outcome 16
Time Frame: Days 0, 28 & 56
Population: Per-Protocol (PP) population that received 2 doses of either vaccine or placebo
Measure: Count of Participants; unit: Participants
Arm/Group | LAIV H7N3: Dose 1 (Day 0) | Placebo: Dose 1 (Day 0) | LAIV H7N3: Day 28 (Dose 2) | Placebo: Day 28 (Dose 2) | LAIV H7N3: Day 56 (28 Days Past Dose 2) | Placebo: Day 56 (28 Days Past Dose 2)
Number analyzed (Participants) | 29 | 10 | 29 | 10 | 29 | 10
Participants
  Positive response | 0 | 0 | 5 | 0 | 5 | 0
  No response | 29 | 10 | 24 | 10 | 24 | 10

ADVERSE EVENTS:
Time Frame: Up to 56 days following dosing
Description: For the assessment of safety, subjects were assessed for adverse reactions twice daily (early morning and late afternoon) for 7 days.
  An ear, nose, and throat (ENT) examination was performed on Days 7, 28, 35, and 56.
  Blood and urine specimens were also collected on Days 7, 28 (prior to administration of the second dose of study vaccine or placebo), 35 and 56, for testing by routine biochemical and hematological blood tests and by urinalysis by dipstick.
Arm/Group | LAIV H7N3: Dose 1 | Placebo: Dose 1 | LAIV H7N3: Dose 2 | Placebo: Dose 2
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/10 | 0/30 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/10 | 0/30 | 0/10
Other Adverse Events (participants affected / at risk) | 20/30 | 5/10 | 25/30 | 8/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LAIV H7N3: Dose 1 (N=30) | Placebo: Dose 1 (N=10) | LAIV H7N3: Dose 2 (N=30) | Placebo: Dose 2 (N=10)
Lymphocytosis (Blood and lymphatic system disorders) | 2 | 0 | 1 | 1
Monocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1
Blood alkaline phosphatase decreased (Investigations) | 0 | 1 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1 | 0
Blood bicarbonate increased (Investigations) | 9 | 3 | 5 | 3
Blood bilirubin increased (Investigations) | 5 | 0 | 2 | 0
Blood calcium increased (Investigations) | 1 | 0 | 3 | 1 (1)
Blood chloride increased (Investigations) | 2 | 1 | 3 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 6 | 0
Eosinophil count increased (Investigations) | 1 | 0 | 1 | 0 (0)
Hemoglobin increased (Investigations) | 1 | 0 | 4 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 2 | 1
Lymphocyte count increased (Investigations) | 6 | 0 | 6 | 1
Mean cell hemoglobin concentration increased (Investigations) | 1 | 0 | 0 | 0
Monocyte count increased (Investigations) | 5 | 0 | 5 | 3
Neutrophil count decreased (Investigations) | 4 | 0 | 5 | 0
White blood cell count increased (Investigations) | 2 | 0 | 2 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 5 | 2
Hemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 | 0 (0)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 1 | 0
Total protein decreased (Investigations) | 0 | 0 | 1 | 0
Red blood cell increased (Investigations) | 0 | 0 | 1 | 0
Red blood cell sedimentation rate increased (Investigations) | 0 | 0 | 2 | 1
Urine leukocyte esterase positive (Investigations) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Study was completed as expected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No